CLINICAL TRIAL: NCT01794520
Title: A Phase 1/2 Study Evaluating the Safety and Pharmacokinetics of ABT-199 in Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: Study Evaluating ABT-199 in Participants With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M13-367; 2012-000589-38 (EudraCT Number)
Expanded Access: NCT03123029 (Available)
Record Dates: First submitted 2012-10-12; First posted 2013-02-20 (Estimated); Results first posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-03

CONDITIONS: Relapsed/Refractory Multiple Myeloma
Keywords: Relapsed multiple myeloma; Refractory multiple myeloma; Multiple myeloma; Relapsed/refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — venetoclax; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- Phase 1: Venetoclax 300 mg (Experimental): Participants in the dose-escalation cohort received 300 mg of venetoclax daily on Days 1 -21 of each cycle after a 2-week lead-in period, during which venetoclax doses were increased weekly.
  Interventions: Drug: Venetoclax
- Phase 1: Venetoclax 600 mg (Experimental): Participants in the dose-escalation cohort received 600 mg of venetoclax daily on Days 1 -21 of each cycle after a 2-week lead-in period, during which venetoclax doses were increased weekly.
  Interventions: Drug: Venetoclax
- Phase 1: Venetoclax 900 mg (Experimental): Participants in the dose-escalation cohort received 900 mg of venetoclax daily on Days 1 -21 of each cycle after a 2-week lead-in period, during which venetoclax doses were increased weekly.
  Interventions: Drug: Venetoclax
- Phase 1: Venetoclax 1200 mg (Experimental): Participants in the dose-escalation cohort received 1200 mg of venetoclax daily on Days 1 -21 of each cycle after a 2-week lead-in period, during which venetoclax doses were increased weekly.
  Interventions: Drug: Venetoclax
- Phase 1 Safety Expansion: Venetoclax 1200 mg (Experimental): Participants in the safety expansion cohort received 1200 mg of venetoclax daily on Days 1 - 21 of each cycle after a 2-week lead-in period, during which venetoclax doses were increased weekly.
  Interventions: Drug: Venetoclax
- Phase 1 Combination: Venetoclax 800 mg/Dexamethasone 20 or 40 mg (Experimental): Participants with t(11;14) translocation multiple myeloma received daily venetoclax at a dose of 800 mg (no lead-in period) on Days 1- 21 of each cycle concomitant with weekly dexamethasone at a dose of 40 mg (20 mg for those aged ≥ 75 years).
  Interventions: Drug: Venetoclax; Drug: Dexamethasone
- Phase 2 Expansion: Venetoclax 800 mg/Dexamethasone 20 or 40 mg (Experimental): The Phase 2 cohort further explored the efficacy of venetoclax in combination with dexamethasone in relapsed or refractory participants with t(11;14) translocation multiple myeloma. Participants received daily venetoclax at a dose of 800 mg (no lead-in period) on Days 1- 21 of each cycle concomitant with weekly dexamethasone at a dose of 40 mg (20 mg for those aged ≥ 75 years).
  Interventions: Drug: Venetoclax; Drug: Dexamethasone

INTERVENTIONS:
Drug: Venetoclax — Each dose of venetoclax was to be taken with approximately 240 mL of water. On days that pre-dose pharmacokinetic (PK) sampling was required, dosing was to occur in the morning at the clinic at approximately 0900 (± 1 hour) to facilitate PK sampling. Dose Escalation cohort participants were to take venetoclax within 30 minutes after the completion of a standard low-fat breakfast with approximately 240 mL of water on Cycle 2 Day 1. On all other dosing days, participants were instructed to take venetoclax orally QD within 30 minutes after the completion of a low-fat breakfast. Tablets were to be swallowed whole and must not have been broken, chewed, or crushed.
  Other Names: ABT-199; VENCLEXTA®
Drug: Dexamethasone — Tablets were administered by mouth per the dexamethasone prescribing information.
  Arms: Phase 1 Combination: Venetoclax 800 mg/Dexamethasone 20 or 40 mg; Phase 2 Expansion: Venetoclax 800 mg/Dexamethasone 20 or 40 mg

SUMMARY:
The Phase 1 primary objectives of this study were to assess the safety profile, characterize pharmacokinetics (PK) and determine the dosing schedule, maximum tolerated dose (MTD), and recommended Phase 2 dose (RPTD) of ABT-199 (venetoclax) when administered in participants with relapsed or refractory multiple myeloma. This study also assessed the safety profile and PK of venetoclax in combination with dexamethasone in participants with t(11;14)-positive multiple myeloma.

The Phase 2 primary objective was to further evaluate the objective response rate (ORR) and very good partial response or better rate (VGPR+) in participants with t(11;14)-positive multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* ECOG (Eastern Cooperative Oncology Group) performance score of 1 or 0. Participants in the Phase 2 portion: ECOG performance score of 2, 1, or 0.
* Diagnosis of multiple myeloma (MM) previously treated with at least one prior line of therapy.

  * Induction therapy followed by stem cell transplant and maintenance therapy will be considered a single line of therapy.
  * For Safety Expansion, participants must have been previously treated with a proteasome inhibitor (e.g., bortezomib) and an immunomodulatory agent (e.g., thalidomide, lenalidomide).
  * For Venetoclax-Dexamethasone Combination, participants must have been previously treated with a proteasome inhibitor (e.g., bortezomib) and an immunomodulatory agent (e.g., thalidomide, lenalidomide) AND have t(11;14)-positive multiple myeloma per the central lab testing.
  * For Phase 2, participants must have MM positive for the t(11;14) translocation, as determined by an analytically validated fluorescence in situ hybridization (FISH) assay per the central laboratory testing (enrollment with local t(11;14)-positive FISH results only will be considered at the discretion of the Therapeutic Area MD). Participants must have evidence of disease progression on or within 60 days of last dose of most recent previous treatment based on International Myeloma Working Group (IMWG) criteria AND must have previously received at least 2 lines of therapy, including an immunomodulatory drug (lenalidomide or pomalidomide), a proteasome inhibitor (bortezomib, carfilzomib or ixazomib), daratumumab, and glucocorticoids.

    * For US participants: Daratumumab combination regimen must be one of the prior lines of therapy (for this study, daratumumab plus corticosteroids will not be considered a combination regimen).
    * For Non-US participants: Either daratumumab monotherapy or combination therapy is acceptable. Daratumumab monotherapy will be limited to approximately 20 percent of the total number of Phase 2 participants.
* Measurable disease at Screening:

  * Serum monoclonal protein of at least 1.0 g/dL (10g/L) by protein electrophoresis.
  * At least 200 mg of monoclonal protein in the urine on 24-hr electrophoresis.
  * Serum immunoglobulin free light chain of at least 10 mg/dL and abnormal serum immunoglobulin kappa to lambda free light chain ratio.
* Participants with a history of autologous or allogenic stem cell transplantation must have adequate peripheral blood counts independent of any growth factor support, and have recovered from any transplant related toxicity(s) and be:

  * At least 100 days post-autologous transplant prior to first dose of study drug or
  * At least 6 months post-allogenic transplant prior to first dose of study drug and not have active graft-versus-host disease (GVHD), i.e., requiring treatment.
* Meet the following laboratory parameters, per the reference range, at least once during the screening period:

  * Absolute Neutrophil Count (ANC) of at least 1000/μL (Participants may use growth factor support to achieve ANC eligibility criteria).
  * Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) not higher than 3 x Upper Limit of Normal Range (ULN).
  * Calculated creatinine clearance of at least 30 mL/min using a modified Cockcroft-Gault calculation.
  * Platelet count of at least 30,000 mm³ (independent of transfusion for 2 weeks).
  * Hemoglobin of at least 8.0 g/dL (participants may receive blood transfusion to achieve hemoglobin eligibility criteria).
  * Total bilirubin not higher than 1.5 x ULN (Participants with Gilbert's Syndrome may have bilirubin higher than 1.5 x ULN).

Exclusion Criteria:

* Exhibits evidence of other clinically significant uncontrolled condition(s), including, but not limited to:

  * Acute infection within 14 days prior to first dose of study drug requiring antibiotic, antifungal, or antiviral therapy.
  * Diagnosis of fever and neutropenia within 1 week prior to first dose of study drug.
* Cardiovascular disability status of New York Heart Association Class ≥ 3.
* Significant history of renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, cardiovascular or hepatic disease, within the last 6 months that, in the opinion of the investigator, would adversely affect his/her participation in the study.
* History of other active malignancies other than multiple myeloma within the past 3 years prior to study entry, with the following exceptions:

  * Adequately treated in situ carcinoma of the cervix uteri;
  * Basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin;
  * Localized prostate cancer Gleason grade 6 or lower AND with stable prostate specific antigen (PSA) levels off treatment
  * Previous malignancy confined and surgically resected (or treated with other modalities) with curative intent.
* Known Human Immunodeficiency Viral (HIV) infection.
* Active hepatitis B or C infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2012-10-10 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2021-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (29):
- United States (21):
  - Mayo Clinic - Scottsdale /ID# 75808, Scottsdale, Arizona
  - University of Arkansas for Medical Sciences /ID# 170002, Little Rock, Arkansas
  - Yale University /ID# 203704, New Haven, Connecticut
  - Emory University, Winship Cancer Institute /ID# 74993, Atlanta, Georgia
  - Ingalls Memorial Hosp /ID# 205346, Harvey, Illinois
  - Tulane Cancer Center Clinic /ID# 204123, New Orleans, Louisiana
  - Tufts Medical Center /ID# 203814, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center Michigan Medicine /ID# 170007, Ann Arbor, Michigan
  - Mayo Clinic - Rochester /ID# 74994, Rochester, Minnesota
  - Hattiesburg Clinic /ID# 201187, Hattiesburg, Mississippi
  - Washington University-School of Medicine /ID# 76094, St Louis, Missouri
  - University of Nebraska Medical Center /ID# 169158, Omaha, Nebraska
  - The John Theurer Cancer /ID# 200248, Hackensack, New Jersey
  - Duke Cancer Center /ID# 129356, Durham, North Carolina
  - University Hospitals - Seidman Cancer Center /ID# 204502, Cleveland, Ohio
  - Ohio State Cancer Center /ID# 200249, Columbus, Ohio
  - Avera Cancer Institute /ID# 204178, Sioux Falls, South Dakota
  - Baylor University Medical Ctr. /ID# 170056, Dallas, Texas
  - Swedish Cancer Institute - Edmonds /ID# 170006, Seattle, Washington
  - Univ of Wisconsin Hosp/Clinics /ID# 200246, Madison, Wisconsin
  - Medical College of Wisconsin /ID# 205229, Milwaukee, Wisconsin
- Belgium (3):
  - UZ Brussel /ID# 170711, Jette, Brussels Capital
  - ZNA Stuivenberg /ID# 170067, Antwerp
  - Duplicate_University Hospital Leuven /ID# 170715, Leuven
- France (4):
  - CHRU Lille - Hopital Claude Huriez /ID# 74995, Lille, Hauts-de-France
  - CHRU Tours - Hopital Bretonneau /ID# 126639, Tours, Indre-et-Loire
  - CHU de Nantes, Hotel Dieu -HME /ID# 75033, Nantes, Pays de la Loire Region
  - Duplicate_CHU Grenoble - Hopital Michallon /ID# 126658, Grenoble
- Ulleval, OUS /ID# 170707, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Badawi M, Coppola S, Eckert D, Gopalakrishnan S, Engelhardt B, Doelger E, Huang W, Dobkowska E, Kumar S, Menon RM, Salem AH. Venetoclax in biomarker-selected multiple myeloma patients: Impact of exposure on clinical efficacy and safety. Hematol Oncol. 2024 Jan;42(1):e3222. doi: 10.1002/hon.3222. Epub 2023 Sep 23. PMID 37740931
- [Derived] Kumar S, Kaufman JL, Gasparetto C, Mikhael J, Vij R, Pegourie B, Benboubker L, Facon T, Amiot M, Moreau P, Punnoose EA, Alzate S, Dunbar M, Xu T, Agarwal SK, Enschede SH, Leverson JD, Ross JA, Maciag PC, Verdugo M, Touzeau C. Efficacy of venetoclax as targeted therapy for relapsed/refractory t(11;14) multiple myeloma. Blood. 2017 Nov 30;130(22):2401-2409. doi: 10.1182/blood-2017-06-788786. Epub 2017 Oct 10. PMID 29018077
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — https://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Intent-to-Treat (ITT) population: all participants who received at least one dose of study drug
Period: Overall Study
Arm/Group | Phase 1: Venetoclax 300 mg | Phase 1: Venetoclax 600 mg | Phase 1: Venetoclax 900 mg | Phase 1: Venetoclax 1200 mg | Phase 1 Safety Expansion: Venetoclax 1200 mg | Phase 1 Combination: Venetoclax 800 mg/Dexamethasone 20 or 40 mg | Phase 2 Expansion: Venetoclax 800 mg/Dexamethasone 20 or 40 mg
Started | 6 | 9 | 6 | 9 | 36 | 20 | 31
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 9 | 6 | 9 | 36 | 20 | 31
Not completed — Adverse events- related to progression | 0 | 0 | 1 | 2 | 0 | 1 | 0
Not completed — Adverse event- not related to progression | 1 | 1 | 0 | 0 | 2 | 0 | 0
Not completed — Progressive disease | 5 | 6 | 2 | 5 | 27 | 18 | 0
Not completed — Withdrew consent | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Toxicity | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Study terminated by sponsor | 0 | 0 | 1 | 0 | 1 | 0 | 7
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0 | 22
Not completed — Other, not specified | 0 | 0 | 1 | 1 | 4 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population: all participants who received at least one dose of study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1: Venetoclax 300 mg | Phase 1: Venetoclax 600 mg | Phase 1: Venetoclax 900 mg | Phase 1: Venetoclax 1200 mg | Phase 1 Safety Expansion: Venetoclax 1200 mg | Phase 1 Combination: Venetoclax 800 mg/Dexamethasone 20 or 40 mg | Phase 2 Expansion: Venetoclax 800 mg/Dexamethasone 20 or 40 mg | Total
Number analyzed (Participants) | 6 | 9 | 6 | 9 | 36 | 20 | 31 | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (7.32) | 63.1 (9.03) | 61.8 (12.06) | 67.3 (8.32) | 60.8 (10.58) | 63.4 (8.13) | 64.9 (8.31) | 63.1 (9.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 5 | 5 | 23 | 3 | 13 | 52
  Male | 5 | 7 | 1 | 4 | 13 | 17 | 18 | 65
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6 | 9 | 4 | 6 | 34 | 17 | 24 | 100
  Black | 0 | 0 | 1 | 1 | 2 | 2 | 5 | 11
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Multi Race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Missing | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study drug. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent adverse events/treatment-emergent serious adverse events (TEAEs/TESAEs) are defined as any event that began or worsened in severity on or after the first dose of study drug.
Time Frame: From first dose of study drug until 30 days following last dose of study drug (up to 2482 days)
Population: Safety population: all participants who received at least one dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Venetoclax 300 mg | Phase 1: Venetoclax 600 mg | Phase 1: Venetoclax 900 mg | Phase 1: Venetoclax 1200 mg | Phase 1 Safety Expansion: Venetoclax 1200 mg | Phase 1 Combination: Venetoclax 800 mg/Dexamethasone 20 or 40 mg | Phase 2 Expansion: Venetoclax 800 mg/Dexamethasone 20 or 40 mg
Number analyzed (Participants) | 6 | 9 | 6 | 9 | 36 | 20 | 31
Participants
  Any TEAE | 6 | 9 | 6 | 9 | 36 | 19 | 30
  TESAE | 1 | 4 | 3 | 3 | 15 | 6 | 16

2. Primary Outcome: Phase 1: Maximum Observed Plasma Concentration (Cmax) of Venetoclax
Description: Cmax is the highest concentration that a drug achieves in the blood after administration in a dosing interval.
Time Frame: Cycle 2, Day 1 at predose, 2, 4, 6, 8, and 24 hours postdose
Population: Phase 1 dose escalation and safety expansion participants with available data
Measure: Mean (Standard Deviation); unit: µg/mL
Groups:
- 300 mg Venetoclax: Participants who received a 300 mg dose of venetoclax administered on the intensive pharmacokinetic sampling day
- 600 mg Venetoclax: Participants who received a 600 mg dose of venetoclax administered on the intensive pharmacokinetic sampling day
- 900 mg Venetoclax: Participants who received a 900 mg dose of venetoclax administered on the intensive pharmacokinetic sampling day
- 1200 mg Venetoclax: Participants who received a 1200 mg dose of venetoclax administered on the intensive pharmacokinetic sampling day
Arm/Group | 300 mg Venetoclax | 600 mg Venetoclax | 900 mg Venetoclax | 1200 mg Venetoclax
Number analyzed (Participants) | 6 | 5 | 4 | 12
µg/mL | 0.897 (0.593) | 2.56 (1.77) | 1.85 (1.30) | 4.16 (1.52)

3. Primary Outcome: Phase 1: Time to Maximum Observed Plasma Concentration (Tmax) of Venetoclax
Description: Tmax is the the time at which the maximum plasma concentration (Cmax) is observed.
Time Frame: Cycle 2, Day 1 at predose, 2, 4, 6, 8, and 24 hours postdose
Population: Phase 1 dose escalation and safety expansion participants with available data
Measure: Median (Full Range); unit: hours
Arm/Group | 300 mg Venetoclax | 600 mg Venetoclax | 900 mg Venetoclax | 1200 mg Venetoclax
Number analyzed (Participants) | 6 | 5 | 4 | 12
hours | 5.0 [2.0 to 8.0] | 8.0 [2.7 to 8.0] | 6.0 [4.0 to 8.0] | 6.1 [4.0 to 8.0]

4. Primary Outcome: Phase 1: Area Under the Plasma Concentration-Time Curve Over Time From 0 to 24 Hours (AUC0-24) of Venetoclax
Description: AUC is a measure of how long and how much drug is present in the body after dosing.
Time Frame: Cycle 2, Day 1 at predose, 2, 4, 6, 8, and 24 hours postdose (dose escalation cohort); (1200 mg dose): Cycle 2, Day 1 at predose (safety expansion cohort, 1200 mg dose)
Population: Phase 1 dose escalation and safety expansion participants with available data
Measure: Mean (Standard Deviation); unit: µg•h/mL
Arm/Group | 300 mg Venetoclax | 600 mg Venetoclax | 900 mg Venetoclax | 1200 mg Venetoclax
Number analyzed (Participants) | 6 | 5 | 3 | 9
µg•h/mL | 13.0 (8.31) | 38.2 (25.1) | 26.3 (20.1) | 71.5 (35.8)

5. Primary Outcome: Phase 2: Overall Response Rate
Description: Overall response rate is defined as the percentage of participants with documented best overall response of Partial Response (PR) or better (PR, Very good partial response [VGPR], Complete response [CR], or Stringent complete response [sCR]) per 2016 standard International Myeloma Working Group (IMWG) criteria.
Time Frame: Response was assessed at Cycle 2, Day 1, and on Day 1 of every cycle thereafter; estimated median time on follow-up was 31.7 months
Population: All enrolled Phase 2 participants who received venetoclax and had active disease at baseline; primary efficacy endpoints were pre-specified for Phase 2 only, and are reported for all participants with available data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2 Expansion: Venetoclax 800 mg/Dexamethasone 20 or 40 mg
Number analyzed (Participants) | 31
percentage of participants | 48.4 [30.2 to 66.9]

6. Primary Outcome: Phase 2: Very Good Partial Response Rate or Better
Description: The percentage of participants with documented best overall response of Very Good Partial Response (VGPR) or better (VGPR, Complete response [CR], or Stringent complete response [sCR]) per 2016 standard International Myeloma Working Group (IMWG) criteria was computed.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2 Expansion: Venetoclax 800 mg/Dexamethasone 20 or 40 mg
Number analyzed (Participants) | 31
percentage of participants | 35.5 [19.2 to 54.6]

7. Secondary Outcome: Phase 1: Overall Response Rate
Description: Overall response rate is defined as the percentage of participants with documented best overall response of Partial Response (PR) or better (PR, Very good partial response [VGPR], Complete response [CR], or Stringent complete response [sCR]) per 2011 International Myeloma Working Group (IMWG) criteria.
Time Frame: Response was assessed at Cycle 2, Day 1, and on Day 1 of every cycle thereafter; estimated median time on follow-up was 8.1 months
Population: All enrolled Phase 1 participants who had active disease at baseline and received venetoclax
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1: Venetoclax 300 mg | Phase 1: Venetoclax 600 mg | Phase 1: Venetoclax 900 mg | Phase 1: Venetoclax 1200 mg | Phase 1 Safety Expansion: Venetoclax 1200 mg | Phase 1 Combination: Venetoclax 800 mg/Dexamethasone 20 or 40 mg
Number analyzed (Participants) | 6 | 9 | 6 | 9 | 36 | 20
percentage of participants | 0 [0.0 to 45.9] | 11.1 [0.3 to 48.2] | 16.7 [0.4 to 64.1] | 0 [0.0 to 33.6] | 36.1 [20.8 to 53.8] | 65.0 [40.8 to 84.6]

8. Secondary Outcome: Time to Response (TTR)
Description: TTR is defined as the number of days from the date of first dose of study drug until the date of their first favorable response of Partial Response (PR) or better (PR, Very good partial response [VGPR], Complete response [CR], or Stringent complete response [sCR]) per 2011 International Myeloma Working Group (IMWG) criteria (Phase 1) or 2016 IMWG criteria (Phase 2). If a participant did not experience a favorable response, they were to be censored at the date of last adequate assessment. TTR was analyzed by Kaplan- Meier (K-M)\ methodology.
Time Frame: Response was assessed at Cycle 2, Day 1, and on Day 1 of every cycle thereafter; Estimated median time on follow-up was 8.1 months for Phase 1 and 31.7 months for Phase 2
Population: All enrolled participants who received venetoclax, had active disease at baseline, and achieved a response (PR or better)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1: Venetoclax 300 mg | Phase 1: Venetoclax 600 mg | Phase 1: Venetoclax 900 mg | Phase 1: Venetoclax 1200 mg | Phase 1 Safety Expansion: Venetoclax 1200 mg | Phase 1 Combination: Venetoclax 800 mg/Dexamethasone 20 or 40 mg | Phase 2 Expansion: Venetoclax 800 mg/Dexamethasone 20 or 40 mg
Number analyzed (Participants) | 0 | 1 | 1 | 0 | 13 | 13 | 15
months |  | NA [1.9 to NA] — Not estimable/calculable due to low number of participants with events | NA [1.2 to NA] — Not estimable/calculable due to low number of participants with events |  | 9.0 [1.9 to NA] — Not estimable/calculable due to low number of participants with events | 2.6 [1.4 to NA] — Not estimable/calculable due to low number of participants with events | 0.8 [0.7 to NA] — Not estimable/calculable due to low number of participants with events

9. Secondary Outcome: Time to Progression (TTP)
Description: TTP is defined as the number of days from the date of first dose of study drug to the date of first documented disease progression or death due to multiple myeloma, whichever occurs first. TTP was analyzed by Kaplan- Meier (K-M) methodology.
Time Frame: Estimated median duration of follow-up was 8.1 months for Phase 1 and 31.7 months for Phase 2
Population: All enrolled participants who received venetoclax
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1: Venetoclax 300 mg | Phase 1: Venetoclax 600 mg | Phase 1: Venetoclax 900 mg | Phase 1: Venetoclax 1200 mg | Phase 1 Safety Expansion: Venetoclax 1200 mg | Phase 1 Combination: Venetoclax 800 mg/Dexamethasone 20 or 40 mg | Phase 2 Expansion: Venetoclax 800 mg/Dexamethasone 20 or 40 mg
Number analyzed (Participants) | 6 | 9 | 6 | 9 | 36 | 20 | 31
months | 5.0 [3.9 to NA] — Not estimable/calculable due to low number of participants with events | 2.0 [0.5 to NA] — Not estimable/calculable due to low number of participants with events | 1.2 [0.4 to NA] — Not estimable/calculable due to low number of participants with events | 1.9 [0.5 to NA] — Not estimable/calculable due to low number of participants with events | 4.2 [1.9 to 10.2] | 12.2 [4.2 to 20.9] | 11.2 [5.2 to 18.4]

10. Secondary Outcome: Duration of Response
Description: DOR is defined as the number of days from the date of first response of Partial Response (PR) or better to the date of first documented disease progression or death due to multiple myeloma, whichever occurs first. DOR was analyzed by Kaplan- Meier (K-M) methodology.
Time Frame: Assessed at Cycle 2, Day 1, and on Day 1 of every cycle thereafter; estimated median duration of follow-up was 8.1 months for Phase 1 and 31.7 months for Phase 2
Population: All enrolled participants who received venetoclax, had active disease at baseline, and achieved a response of PR or better
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1: Venetoclax 300 mg | Phase 1: Venetoclax 600 mg | Phase 1: Venetoclax 900 mg | Phase 1: Venetoclax 1200 mg | Phase 1 Safety Expansion: Venetoclax 1200 mg | Phase 1 Combination: Venetoclax 800 mg/Dexamethasone 20 or 40 mg | Phase 2 Expansion: Venetoclax 800 mg/Dexamethasone 20 or 40 mg
Number analyzed (Participants) | 0 | 1 | 1 | 0 | 13 | 13 | 15
months |  | 9.7 [NA to NA] — Not estimable/calculable due to low number of participants with events | NA [NA to NA] — Not estimable/calculable due to low number of participants with events |  | 17.3 [7.8 to 27.0] | 13.1 [5.7 to 21.9] | 17.5 [7.6 to 28.8]

11. Secondary Outcome: Phase 2: Progression-Free Survival (PFS)
Description: PFS is defined as the number of days from the date of the first dose of study treatment to the date of first documented disease progression or death due to any cause, whichever occurs first. PFS was analyzed by Kaplan-Meier methodology.
Time Frame: Estimated median duration of follow-up was 31.7 months
Population: All enrolled Phase 2 participants who received venetoclax and had active disease at baseline; this endpoint was pre-specified for Phase 2 only, data are reported for all participants with available data
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2 Expansion: Venetoclax 800 mg/Dexamethasone 20 or 40 mg
Number analyzed (Participants) | 31
months | 11.2 [5.2 to 18.4]

12. Secondary Outcome: Phase 2: Overall Survival (OS)
Description: OS is defined as the number of days from the date of the first dose of study drug to the date of death due to any cause. If a participant was not known to have died, OS was censored at the last known alive date. The distribution of OS was estimated using Kaplan-Meier methodology.
Time Frame: Estimated median duration of follow-up was 31.7 months
Population: All enrolled Phase 2 participants who received venetoclax; this endpoint was pre-specified for Phase 2 only, data are reported for all participants with available data
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2 Expansion: Venetoclax 800 mg/Dexamethasone 20 or 40 mg
Number analyzed (Participants) | 31
months | 18.4 [8.2 to 24.3]

13. Secondary Outcome: Phase 2: Mean Change From Baseline in Brief Pain Inventory - Short Form (BPI-SF) Worst Pain
Description: The BPI-SF is a pain-specific measure developed to assess patient-reported severity (or intensity) of pain (4 items) and the impact of pain on daily functioning (7 items) in patients with cancer pain. The four pain severity items assess pain at its "worst in last 24 hours," "least in last 24 hours," "average," and "now" (current pain). For these items, participants are asked to rate their pain on an 11-point numeric rating scale with anchors of 0 (no pain) and 10 (pain as bad as you can imagine). The Worst Pain scores range from 0 to 10, with higher scores indicating severe pain. Negative changes from baseline indicate improvement.
Time Frame: Baseline; Cycle 3, Day 1; Cycle 5, Day 1; Cycle 7, Day 1; Cycle 9, Day 1; Cycle 11, Day 1; Cycle 13, Day 1; Cycle 15, Day 1; Cycle 17, Day 1; Cycle 19, Day 1; Cycle 21, Day 1; Cycle 23, Day 1; Cycle 25, Day 1; Final visit
Population: Intent-to-Treat (ITT) population: all participants who received at least one dose of study drug; participants who have both baseline and post-baseline values are included in the analysis at each visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phase 2 Expansion: Venetoclax 800 mg/Dexamethasone 20 or 40 mg
Number analyzed (Participants) | 16
units on a scale
  Cycle 3, Day 1 | 0.2 (2.47)
  Cycle 5, Day 1: number analyzed (Participants) | 10
  Cycle 5, Day 1 | -0.9 (1.43)
  Cycle 7, Day 1: number analyzed (Participants) | 8
  Cycle 7, Day 1 | -0.9 (1.20)
  Cycle 9, Day 1: number analyzed (Participants) | 8
  Cycle 9, Day 1 | -0.9 (1.46)
  Cycle 11, Day 1: number analyzed (Participants) | 7
  Cycle 11, Day 1 | -1.1 (1.62)
  Cycle 13, Day 1: number analyzed (Participants) | 7
  Cycle 13, Day 1 | 0.5 (3.84)
  Cycle 15, Day 1: number analyzed (Participants) | 7
  Cycle 15, Day 1 | -0.6 (1.27)
  Cycle 17, Day 1: number analyzed (Participants) | 6
  Cycle 17, Day 1 | -1.6 (1.29)
  Cycle 19, Day 1: number analyzed (Participants) | 3
  Cycle 19, Day 1 | -1.8 (2.00)
  Cycle 21, Day 1: number analyzed (Participants) | 2
  Cycle 21, Day 1 | -1.6 (2.30)
  Cycle 23, Day 1: number analyzed (Participants) | 2
  Cycle 23, Day 1 | -1.6 (2.30)
  Cycle 25, Day 1: number analyzed (Participants) | 1
  Cycle 25, Day 1 | -3.8
  Final visit | -0.3 (1.86)

14. Secondary Outcome: Phase 2: Mean Change From Baseline in Physical Functioning Scale of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30)
Description: The QLQ-C30 is a 30-item subject self-report questionnaire composed of both multi-item and single scales, including five functional scales (physical, role, emotional, social, and cognitive), three symptom scales (fatigue, nausea and vomiting, and pain), a global health status/quality of life scale, and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). For the Physical Functioning scale, participants rate five items on a four-point scale, with 1 as "not at all" and 4 as "very much." The Physical Functioning Scale scores range from 0 to 100 and were calculated per the EORTC QLQ-C30 Scoring Manual (3rd edition), version 3.0. A high scale score represents high/healthy level of functioning. Positive changes from baseline indicate improvement.
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phase 2 Expansion: Venetoclax 800 mg/Dexamethasone 20 or 40 mg
Number analyzed (Participants) | 16
units on a scale
  Cycle 3, Day 1 | -3.7 (21.90)
  Cycle 5, Day 1: number analyzed (Participants) | 10
  Cycle 5, Day 1 | 4.0 (15.78)
  Cycle 7, Day 1: number analyzed (Participants) | 8
  Cycle 7, Day 1 | 8.3 (11.13)
  Cycle 9, Day 1: number analyzed (Participants) | 8
  Cycle 9, Day 1 | 8.3 (11.13)
  Cycle 11, Day 1: number analyzed (Participants) | 7
  Cycle 11, Day 1 | 15.2 (9.97)
  Cycle 13, Day 1: number analyzed (Participants) | 7
  Cycle 13, Day 1 | 11.4 (14.76)
  Cycle 15, Day 1: number analyzed (Participants) | 7
  Cycle 15, Day 1 | 14.3 (11.17)
  Cycle 17, Day 1: number analyzed (Participants) | 6
  Cycle 17, Day 1 | 8.9 (13.11)
  Cycle 19, Day 1: number analyzed (Participants) | 3
  Cycle 19, Day 1 | -0.0 (11.55)
  Cycle 21, Day 1: number analyzed (Participants) | 2
  Cycle 21, Day 1 | -13.3 (28.28)
  Cycle 23, Day 1: number analyzed (Participants) | 2
  Cycle 23, Day 1 | -3.3 (14.14)
  Cycle 25, Day 1: number analyzed (Participants) | 1
  Cycle 25, Day 1 | 6.7
  Final visit | -5.0 (19.40)

15. Secondary Outcome: Phase 2: Mean Change From Baseline in Global Health Status/Quality of Life Scale of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30)
Description: The QLQ-C30 is a 30-item subject self-report questionnaire composed of both multi-item and single scales, including five functional scales (physical, role, emotional, social, and cognitive), three symptom scales (fatigue, nausea and vomiting, and pain), a global health status/quality of life scale, and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). For the Global Health Status/Quality of Life scale, participants rate two items on a seven point scale, with 1 as "very poor" and 7 as "excellent." The Global Health Status/Quality of Life scale ranges from 0 to 100 and was calculated per the EORTC QLQ-C30 Scoring Manual (3rd edition), version 3.0. A high score for the global health status/QoL represents a high QoL. Positive changes from baseline indicate improvement.
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phase 2 Expansion: Venetoclax 800 mg/Dexamethasone 20 or 40 mg
Number analyzed (Participants) | 16
units on a scale
  Cycle 3, Day 1 | -5.2 (25.44)
  Cycle 5, Day 1: number analyzed (Participants) | 10
  Cycle 5, Day 1 | 6.7 (5.27)
  Cycle 7, Day 1: number analyzed (Participants) | 8
  Cycle 7, Day 1 | 3.1 (7.63)
  Cycle 9, Day 1: number analyzed (Participants) | 8
  Cycle 9, Day 1 | 8.3 (11.79)
  Cycle 11, Day 1: number analyzed (Participants) | 7
  Cycle 11, Day 1 | 0.0 (11.79)
  Cycle 13, Day 1: number analyzed (Participants) | 7
  Cycle 13, Day 1 | -6.0 (6.30)
  Cycle 15, Day 1: number analyzed (Participants) | 7
  Cycle 15, Day 1 | 4.8 (8.13)
  Cycle 17, Day 1: number analyzed (Participants) | 6
  Cycle 17, Day 1 | -1.4 (12.27)
  Cycle 19, Day 1: number analyzed (Participants) | 3
  Cycle 19, Day 1 | -19.4 (4.81)
  Cycle 21, Day 1: number analyzed (Participants) | 2
  Cycle 21, Day 1 | -33.3 (23.57)
  Cycle 23, Day 1: number analyzed (Participants) | 2
  Cycle 23, Day 1 | -8.3 (0.00)
  Cycle 25, Day 1: number analyzed (Participants) | 1
  Cycle 25, Day 1 | -8.3
  Final visit | -11.5 (23.55)

16. Secondary Outcome: Phase 2: Mean Change From Baseline in Patient Reported Outcomes Measurement Information System [PROMIS] Cancer Fatigue Short Form [SF] Score
Description: PROMIS Cancer Fatigue SF is a seven item questionnaire that assesses the impact and experience of fatigue over the past 7 days. All questions employ the following five response options: 1 = Not at all, 2 = A little bit, 3 = Somewhat, 4 = Quite a bit, and 5 = Very much. The total raw score is the sum of the responses to each question and is converted to a T-score. The T-score re-scales the total raw score to a standardized score with a mean of 50 and a standard deviation of 10. The [PROMIS] Cancer Fatigue Short Form [SF] 7a T-Scores range from 29.4 to 83.2, with higher scores indicating more fatigue. Negative changes from baseline indicate improvement.
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Phase 2 Expansion: Venetoclax 800 mg/Dexamethasone 20 or 40 mg
Number analyzed (Participants) | 16
T-score
  Cycle 3, Day 1 | 0.6 (5.88)
  Cycle 5, Day 1: number analyzed (Participants) | 10
  Cycle 5, Day 1 | -2.9 (5.30)
  Cycle 7, Day 1: number analyzed (Participants) | 8
  Cycle 7, Day 1 | -1.8 (4.21)
  Cycle 9, Day 1: number analyzed (Participants) | 8
  Cycle 9, Day 1 | -1.6 (4.85)
  Cycle 11, Day 1: number analyzed (Participants) | 7
  Cycle 11, Day 1 | 0.1 (7.24)
  Cycle 13, Day 1: number analyzed (Participants) | 7
  Cycle 13, Day 1 | 1.0 (4.54)
  Cycle 15, Day 1: number analyzed (Participants) | 7
  Cycle 15, Day 1 | -3.4 (5.69)
  Cycle 17, Day 1: number analyzed (Participants) | 6
  Cycle 17, Day 1 | 0.6 (7.36)
  Cycle 19, Day 1: number analyzed (Participants) | 3
  Cycle 19, Day 1 | 6.6 (2.25)
  Cycle 21, Day 1: number analyzed (Participants) | 2
  Cycle 21, Day 1 | 11.6 (6.51)
  Cycle 23, Day 1: number analyzed (Participants) | 2
  Cycle 23, Day 1 | 6.0 (0.57)
  Cycle 25, Day 1: number analyzed (Participants) | 1
  Cycle 25, Day 1 | 5.6
  Final visit | 1.4 (6.51)

ADVERSE EVENTS:
Time Frame: All-cause mortality is reported from enrollment to end of study; median time on follow up was 6.6, 3.4, 3.8, 3.0, 11.0, 13.2, and 31.7 months for Phase 1 300 mg Ven, Phase 1 600 mg Ven, Phase 1 900 mg Ven, Phase 1 1200 mg Ven, Phase 1 Safety Expansion Ven 1200 mg, Phase 1 Combination Ven 800 mg/Dex, and Phase 2 Expansion Ven 800 mg/Dex, respectively.
Description: TEAEs and SAEs were collected from first dose of study drug until 30 days after last dose of study drug; mean duration on study drug was 171.8, 283.1, 474.5, 76.4, 315.4, 400.0, and 240.3 days for Phase 1 300 mg Ven, Phase 1 600 mg Ven, Phase 1 900 mg Ven, Phase 1 1200 mg Ven, Phase 1 Safety Expansion Ven 1200 mg, Phase 1 Combination Ven 800 mg/Dex, and Phase 2 Expansion Ven 800 mg/Dex, respectively.
Arm/Group | Phase 1: Venetoclax 300 mg | Phase 1: Venetoclax 600 mg | Phase 1: Venetoclax 900 mg | Phase 1: Venetoclax 1200 mg | Phase 1 Safety Expansion: Venetoclax 1200 mg | Phase 1 Combination: Venetoclax 800 mg/Dexamethasone 20 or 40 mg | Phase 2 Expansion: Venetoclax 800 mg/Dexamethasone 20 or 40 mg
All-Cause Mortality (participants affected / at risk) | 1/6 | 1/9 | 1/6 | 0/9 | 6/36 | 1/20 | 22/31
Serious Adverse Events (participants affected / at risk) | 1/6 | 4/9 | 3/6 | 3/9 | 15/36 | 6/20 | 16/31
Other Adverse Events (participants affected / at risk) | 6/6 | 9/9 | 6/6 | 9/9 | 35/36 | 19/20 | 27/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Venetoclax 300 mg (N=6) | Phase 1: Venetoclax 600 mg (N=9) | Phase 1: Venetoclax 900 mg (N=6) | Phase 1: Venetoclax 1200 mg (N=9) | Phase 1 Safety Expansion: Venetoclax 1200 mg (N=36) | Phase 1 Combination: Venetoclax 800 mg/Dexamethasone 20 or 40 mg (N=20) | Phase 2 Expansion: Venetoclax 800 mg/Dexamethasone 20 or 40 mg (N=31)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
HYPERVISCOSITY SYNDROME (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OESOPHAGITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
CHEST DISCOMFORT (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PAIN (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ANAPHYLACTIC REACTION (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABSCESS BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABSCESS INTESTINAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CANDIDA INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
ENTEROBACTER SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ENTEROCOCCAL SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ENTEROVIRUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ESCHERICHIA SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LISTERIA SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LOCALISED INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PARAINFLUENZAE VIRUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 6 (7) | 0 (0) | 1 (2)
PNEUMONIA ASPIRATION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA INFLUENZAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA KLEBSIELLA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA STREPTOCOCCAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RHINOVIRUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (4)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
STREPTOCOCCAL SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHRONIC MYELOMONOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 2 (2)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SCIATICA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Venetoclax 300 mg (N=6) | Phase 1: Venetoclax 600 mg (N=9) | Phase 1: Venetoclax 900 mg (N=6) | Phase 1: Venetoclax 1200 mg (N=9) | Phase 1 Safety Expansion: Venetoclax 1200 mg (N=36) | Phase 1 Combination: Venetoclax 800 mg/Dexamethasone 20 or 40 mg (N=20) | Phase 2 Expansion: Venetoclax 800 mg/Dexamethasone 20 or 40 mg (N=31)
ANAEMIA (Blood and lymphatic system disorders) | 1 (2) | 3 (3) | 1 (1) | 3 (3) | 5 (5) | 2 (2) | 7 (9)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (5)
LYMPHOPENIA (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 3 (7)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 4 (6) | 1 (2) | 0 (0) | 4 (5) | 1 (1) | 1 (4)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
SINUS TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
EAR PAIN (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
CATARACT (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EYE DISCHARGE (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
EYE PAIN (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
VISUAL ACUITY REDUCED (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 1 (1)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 5 (5) | 1 (1) | 4 (4)
DENTAL CARIES (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 2 (2) | 4 (5) | 2 (5) | 5 (5) | 13 (16) | 7 (8) | 12 (16)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FLATULENCE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
HAEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
MOUTH ULCERATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 6 (7) | 3 (3) | 5 (5) | 18 (23) | 5 (5) | 10 (13)
ODYNOPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PARAESTHESIA ORAL (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
TRICHOGLOSSIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
UMBILICAL HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 4 (6) | 2 (2) | 2 (2) | 4 (5) | 2 (3) | 5 (7)
ASTHENIA (General disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
CHILLS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 0 (0)
FACE OEDEMA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 2 (3) | 1 (1) | 0 (0) | 2 (2) | 15 (16) | 2 (2) | 9 (14)
FEELING COLD (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GAIT DISTURBANCE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
MALAISE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OEDEMA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 4 (5) | 4 (4)
PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
PYREXIA (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 4 (4) | 0 (0)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
BRONCHITIS VIRAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CONJUNCTIVITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
CYSTITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FUNGAL SKIN INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
LOCALISED INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 3 (4) | 1 (2) | 1 (1)
ORAL CANDIDIASIS (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTITIS MEDIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
PARAINFLUENZAE VIRUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
RHINITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
RHINOVIRUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
SINUSITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
SKIN INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TOOTH INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 8 (13) | 6 (11) | 3 (4)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (5) | 0 (0) | 1 (1)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
DENTAL RESTORATION FAILURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HEAD INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
TONGUE INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACTIVATED PARTIAL THROMBOPLASTIN TIME ABNORMAL (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 3 (4) | 1 (4) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 3 (4) | 2 (3)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 2 (2) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 5 (7) | 4 (4) | 4 (4)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 4 (5) | 4 (6)
BLOOD PHOSPHORUS INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
BLOOD THYROID STIMULATING HORMONE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CARDIAC MURMUR (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTRAOCULAR PRESSURE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LIPASE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LYMPHOCYTE COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 9 (13) | 4 (7) | 10 (11)
NEUTROPHIL COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 12 (20) | 3 (5) | 3 (7)
PLATELET COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (2) | 3 (8) | 11 (15) | 3 (5) | 2 (2)
WEIGHT DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 13 (21) | 5 (7) | 1 (3)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 1 (2) | 1 (1) | 1 (3) | 2 (2) | 3 (3)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 2 (2)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 4 (4) | 6 (9) | 6 (6)
HYPERMAGNESAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (4) | 3 (3)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (2)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 6 (6) | 3 (4) | 4 (4)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 9 (11) | 4 (6) | 4 (7)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (5) | 1 (1) | 3 (5)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 3 (3)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 6 (9) | 8 (14) | 3 (4)
MALNUTRITION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
STEROID DIABETES (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 1 (2) | 1 (1) | 6 (9) | 5 (7) | 4 (5)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 7 (7) | 1 (1) | 0 (0)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 1 (1) | 2 (2)
EXOSTOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 1 (1) | 1 (1)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 2 (2) | 3 (3)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 3 (3) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
OSTEONECROSIS OF JAW (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 3 (4)
SPINAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
TENDONITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PANCREATIC NEUROENDOCRINE TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COGNITIVE DISORDER (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 1 (2) | 0 (0) | 3 (3) | 0 (0) | 4 (6) | 1 (1) | 4 (4)
DYSAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HEAD DISCOMFORT (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 10 (13) | 3 (5) | 1 (1)
HEMIPARESIS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPERSOMNIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (5)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
PRESYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
SEIZURE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
SOMNOLENCE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
AGITATION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
INSOMNIA (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 8 (10) | 6 (6)
MOOD ALTERED (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
POLLAKIURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
PROTEINURIA (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
PELVIC PAIN (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (3) | 0 (0) | 0 (0) | 8 (8) | 5 (6) | 5 (7)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 1 (1) | 2 (2) | 0 (0) | 5 (8) | 1 (1) | 5 (6)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 2 (3)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 5 (7) | 2 (3)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 5 (5) | 3 (3)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 3 (4) | 3 (3)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
SNEEZING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
UPPER-AIRWAY COUGH SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ACTINIC KERATOSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
HYPERKERATOSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PAPULE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
PURPURA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 4 (5) | 1 (1) | 1 (2)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
SKIN ATROPHY (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SKIN LESION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
URTICARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
EMBOLISM (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HOT FLUSH (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 2 (2)
HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2021-02-17): https://cdn.clinicaltrials.gov/large-docs/20/NCT01794520/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-11): https://cdn.clinicaltrials.gov/large-docs/20/NCT01794520/SAP_001.pdf